CLINICAL TRIAL: NCT05994196
Title: Evaluation of a Patient Prioritization Software for the Secondary Prioritization of Patients in the Pediatric Emergency Department
Brief Title: Evaluation of a Software for the Secondary Prioritization of Patients in the Pediatric Emergency Department
Acronym: OPTIMUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NI2021_01
Record Dates: First submitted 2023-07-31; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Length of Stay
Keywords: Patient flow; Patient prioritization; Pediatric Emergency Department; Usage assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimum (Experimental): the secondary prioritization software of patients
  Interventions: Behavioral: Optimum, a secondary prioritization software of patients in the pediatric emergency department (ED)
- Control (No Intervention): the standard dashboard of patients

INTERVENTIONS:
Behavioral: Optimum, a secondary prioritization software of patients in the pediatric emergency department (ED) — Optimum®'s purpose is to remove the mental load of prioritization from the Pediatric ED staff. The software first prioritizes the triage of new patients by the ED staff and the first evaluation of a new patient by the medical team. Optimum® then prioritizes blood sample collections and care (for nurses) and checks on imaging results, blood test results or an evaluation by a specialist (for physicians). Lastly, Optimum® prioritizes the final step in patient management by a senior physician, when appropriate.
  Arms: Optimum

SUMMARY:
The goal of this randomized, controlled, open-label trial is to test the use of secondary prioritization software (Optimum®) in the pediatric emergency department (PED).

The aim of this study is to determine:

1. whether the use of this secondary prioritization software (Optimum®) reduces the patients' median length of stay (LOS) in the PED
2. how this software is accepted by the staff. The PED staff will be asked to manage the patients according to the Optimum® software indications (intervention) or according to the standard dashboard (control).

DETAILED DESCRIPTION:
Design: randomized, controlled open-label trial in the PED at Lille University Medical Center, Lille, France.

Period: between March 15th and April 23rd, 2021.

Randomization: each day was randomized for the use of Optimum® software (intervention group) or the PED's standard patient management dashboard (control group).

Inclusion criteria:

- All children admitted between 10:00 am and 0:00 am at the PED.

Exclusion criteria:

* Patients who left without being seen
* Patients admitted to a short-stay unit at the PED.

Authorizations: the study protocol was registered with the French National Data Protection Commission (Commission Nationale de l'Informatique et des Libertés, Paris, France; registration number: DEC21-056). This research was submitted to the institutional review board, which replied that this type of study, without patient intervention, did not require validation by the ethics committee. The patients and their parents were shown a study information sheet at the PED reception desk and were free to object to their child's participation.

The prioritization software: Optimum® was developed in 2015. Five variables with a statistically significant influence on the LOS were identified; the reason for admission, the number of patients present in the PED simultaneously, the prescription of imaging, the prescription of blood tests, and the prescription of treatment. Optimum®'s purpose is to remove the mental load of prioritization from the PED staff. The software first prioritizes the triage of new patients by the PED staff and the first evaluation of a new patient by the medical team. Optimum® then prioritizes blood sample collections and care (for nurses) and checks on imaging results, blood test results or an evaluation by a specialist (for physicians). Lastly, Optimum® prioritizes the final step in patient management by a senior physician, when appropriate.

Primary endpoint: the LOS for each patient. Number of patients needed: with a hypothesis of a 15-minute difference in the LOS between the Optimum® and control groups, when considering a mean of 78 patients/day and a median LOS of 190 minutes, with an α-risk of 0.05 and a power (1-ß risk) of 0.8, a total of 1542 patients had to be included (i.e., 771 per group).

Secondary endpoints:

* number of patients present at the same time in the PED,
* time intervals between each stage in patient management from nurse triage to discharge,
* PED staff's level of satisfaction using the standardized System Usability Scale (SUS).

Study procedures :

1. training of all the PED staff members in use of Optimum® 2 weeks prior to the study.
2. study setting up: with days randomized to Optimum® vs. the standard dashboard using the "random" formula in Excel® (Microsoft Corporation, Redmond, WA, USA). Weekdays and weekend/public holiday days were randomized separately. An investigator not involved in the management of the patients during the study period was present throughout the inclusion period and prospectively recorded the time intervals for each patient's stay in the PED: time of arrival at the PED, evaluation by the triage nurse, the first medical evaluation (by a medical student or a junior physician), the first evaluation by a senior physician, the evaluation by a specialist physician (if applicable), the results of imaging and lab tests (if prescribed), the final medical decision, and discharge.

Data collected: in addition to the LOS and to the time intervals of the different phases of management, the other variables recorded were age, gender, reason for admission, triage level, and mode of discharge. There were five categories of reasons for admission: fever, a respiratory disorder, a digestive tract disorder, trauma, and other reasons.

3) the PED staff involved in the study will fill out the standardized SUS questionnaire as a guide to the perceived utility of the Optimum® software and the level of user satisfaction. According to the literature, the SUS score is considered to be very poor if it is less than 51, poor if between 51 and 68, average if 68, good if between 68 and 80.3, and excellent if greater than 80.3.

Statistical analysis:

1. description of patients' characteristics
2. the normality of the data distributions was checked graphically and using the Shapiro-Wilk test.
3. Intergroup comparisons of the total LOS and the various time intervals during patient management times were performed by covariance analysis.
4. Analysis of the standardized System Usability Scale (SUS) questionnaire filled out by the PED staff at th end of the study to perceive the utility of the Optimum® software and the level of user satisfaction. A Spearman's test was used to analyze the correlation between the age of the PED staff and the SUS score.

ELIGIBILITY:
Inclusion Criteria:

* All children admitted between 10:00 am and 0:00 am

Exclusion Criteria:

* Patients who left without being seen
* Patients subsequently admitted to the short-stay unit

Ages: 3 Days to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1599 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Length of stay | from admission to discharge, assessed up to 1 day.
  the length of stay for each patient

SECONDARY OUTCOMES:
Number of patients present | 1 day
  Number of patients present at the same time in the pediatric emergency department during the study period
Time intervals between each stage | 1 day
  The time intervals between each stage in patient management from nurse triage to discharge
Pediatric emergency department staff satisfaction | through study completion, an average of 3 months
  To measure the pediatric emergency department staff's level of satisfaction with the System Usability Scale. Values range from 0 to 100 points. Higher scores mean a better satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: François Dubos, MD, PhD, Principal Investigator — Lille University Hospital
Locations (1):
- Hôpital Roger Salengro, CHU, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schiro J, Marcilly R, Leroy N, Wawrzyniak C, Martinot A, Pelayo S. Design and evaluation of a patient website to reduce crowding in emergency departments: a preliminary study. Stud Health Technol Inform. 2015;210:663-5. PMID 25991232
- [Background] Windal F, Jeribi K, Ficheur G, Degoul S, Martinot A, Beuscart R, Renard JM. Pediatric emergency department crowding: survival tree clustering for length of patient stay. Stud Health Technol Inform. 2014;205:1095-9. PMID 25160358
- [Background] Gravel J, Fitzpatrick E, Gouin S, Millar K, Curtis S, Joubert G, Boutis K, Guimont C, Goldman RD, Dubrovsky AS, Porter R, Beer D, Doan Q, Osmond MH. Performance of the Canadian Triage and Acuity Scale for children: a multicenter database study. Ann Emerg Med. 2013 Jan;61(1):27-32.e3. doi: 10.1016/j.annemergmed.2012.05.024. Epub 2012 Jul 27. PMID 22841173
- [Derived] Lun T, Schiro J, Cailliau E, Tchokokam J, Liber M, de Jorna C, Martinot A, Dubos F. Randomized controlled open-label trial to evaluate prioritization software for the secondary triage of patients in the pediatric emergency department. Int J Emerg Med. 2024 Apr 8;17(1):53. doi: 10.1186/s12245-024-00623-3. PMID 38589780
- See also: Description of the standardized System Usability Scale (SUS) — https://digital.ahrq.gov/sites/default/files/docs/survey/systemusabilityscale%2528sus%2529_comp%255B1%255D.pdf